CLINICAL TRIAL: NCT03583541
Title: Kyaterekera Project: A Combination Intervention Addressing Sexual Risk-Taking Behaviors Among Vulnerable Women in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Columbia University (Other); Indiana University (Other); Rakai Health Sciences Program (Other); Reach the Youth Uganda (Other)
Responsible Party: Principal Investigator, Fred Ssewamala, William E. Gordon Distinguished Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH116768 (NIH)
Record Dates: First submitted 2018-05-31; First posted 2018-07-11 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Control arm_Bolstered Care; Treatment arm_HIVRR+S+FL; Treatment arm_HIVRR+S+FL+M
Keywords: Vulnerable women; Female sex workers; Combination interventions; Economic empowerment; HIV/AIDS; Sexually transmitted infections; Sub-Saharan Africa; Uganda
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm: Bolstered treatment (Experimental): Women in the control condition (and in the treatment arms) will receive treatment as usual (TAU) for FSW in the study area. Provided by RHSP, TAU includes: health education, HIV testing services, STI screening and treatment in a session that lasts about 2 hours, provided on a quarterly basis. This will be bolstered with 4 sessions provided twice per week for 2 weeks of an evidence-based, HIV/STI risk reduction intervention
  Interventions: Behavioral: HIV Risk Reduction
- Treatment arm: HIVRR+S+FL (Experimental): Women in this arm will receive TAU for FSW and the 4 HIVRR sessions (described above) and a single session following HIVRR specifically describing bank account opening, the matching process, and how to interact with banks. In this session our partnering banks will open up matched savings accounts for women in the two treatment arms. Women in both arms will save money in their matched savings accounts over a 10-month period post HIVRR. The study team will monitor the accounts using the statements received directly from the banks holding the accounts. Participants will receive monthly bank statements indicating their own savings and the associated match (1:1 match rate). They will also receive 6 financial literacy (FL) sessions provided twice a week for 3 weeks
  Interventions: Behavioral: HIV Risk Reduction; Behavioral: Financial Literacy; Behavioral: Matched savings individual development account
- Treatment arm: HIVRR+S+FLM (Experimental): Women in this arm will receive TAU and the 4 HIVRR sessions (as above). Next, they will receive the savings session (described above) and 6 financial literacy (FL) sessions provided twice a week for 3 weeks, followed by 8 mentorship (M) sessions supporting transition to vocational, educational training, employment or business development, and receipt of a matched savings account to be used on short-term and/or long term consumption and skills development per participants own discretion/choice.
  *Revision note: Following COVID-19, with approval from NIMH (on record if requested), the HIVRR+S+FLM treatment arm of the study has been combined with the HIVRR+S+FL treatment arm. The total sample size has been revised to 542 participants, with approval from NIMH.
  Interventions: Behavioral: HIV Risk Reduction; Behavioral: Financial Literacy; Behavioral: Mentorship; Behavioral: Matched savings individual development account

INTERVENTIONS:
Behavioral: HIV Risk Reduction — This is an intervention comprised of 4 sessions provided twice per week for 2 weeks of an evidence-based, HIV/STI risk reduction intervention.
Behavioral: Financial Literacy — This evidence-based Financial Education Core Curriculum addresses the importance of savings, banking services, budgeting debt management. Undarga adaptation for FSWs included shortening and simplifying sessions while retaining core elements; adding weekly check-ins due to safety concerns FSWs share related to intervention participation, and safety planning as needed. We will further adapt sessions in months 1-6 to assure language and illustrative examples are culturally consonant, and to infuse BE principles consistent with HIVRR. During sessions 1 & 2 we will include information on delay discounting, for example, learning to understand the tendency to prefer small immediate rewards over larger available at a later time; sessions 3 & 4 will include details on economic utility; sessions 5 will contain information on salience (e.g. understanding occasions when women may minimize triggers to unsafe sex); and session 6 will address loss aversion.
  Arms: Treatment arm: HIVRR+S+FL; Treatment arm: HIVRR+S+FLM
Behavioral: Mentorship — Mentorship. Mentorship to bridge the transition from FL and savings to a vocational change is a critical component of this intervention. These sessions are intended to support the transition -equipped with financial literacy and savings -to vocational, educational, employment or small business development training using matched savings. The mentorship sessions are adapted from the pilot study and integrate components (e.g., referral and linkage, coaching, exchange visits to model farmers) from income-generating activities provided by our collaborating partner, RTY. All sessions include check-in and individual attention. The first 4 sessions focus on identifying options for vocational, educational, employment or business development training. The second 4 sessions include invited experts in identified areas of interest by group members for more intensive time and attention to individualized needs to make the transition.
  Arms: Treatment arm: HIVRR+S+FLM
Behavioral: Matched savings individual development account — A matched savings individual development account (hereafter IDA) is a savings account held at a local bank whereby deposits made by the woman are matched by the intervention to encourage savings and investment in skills and asset development. The accounts introduce women to financial management skills, introduce them to formal financial institutions, and by matching their deposits, incentivize women to save small amounts. Each woman will receive an IDA held in her own name. Women will be allowed and indeed encouraged to contribute up to 50,000 shillings (~15 USD) per month towards their IDAs. The maximum amount of women's contribution to be matched will be an equivalent of US$15 per month for 10 months. During the intervention, monthly account statements will be generated for women to note their accumulated savings. During the intervention, women will have direct access to both their personal savings deposited in the accounts and the match provided by the study.
  Arms: Treatment arm: HIVRR+S+FL; Treatment arm: HIVRR+S+FLM

SUMMARY:
Guided by Social Cognitive and Asset theories as well as Behavioral Economics (BE) principles,the proposed RCT is carefully designed to test the additive contributions of savings-led microfinance beyond traditional HIV risk reduction (HIVRR) alone in decreasing biologically confirmed STIs, including HIV, improving high risk behavioral outcomes, while concurrently reducing income from sex work. Working within established health care- and outreach-based settings, we will randomly assign 990 FSWs to one of three study arms (11 town centers each): (1) a control arm comprising treatment as usual (TAU) for FSWs (quarterly 2-3 hour health education sessions, HIV testing services, and STI screening), bolstered with 4 evidence-based sessions of HIVRR provided by local providers (n=330 ); or (2) a treatment arm including TAU, 4 sessions of HIVRR, combined with receipt of a matched savings account (HIVRR+S) to be used on short-term and/or long term consumption and skills development per a participant's discretion/choice (n=330); or (3) a treatment arm including TAU, 4 sessions of HIVRR, combined with a matched savings account for short-term and/or long term consumption and skills development, plus 6 sessions of financial literacy with integrated BE principles (e.g., delay discounting, economic utility, information salience, and loss aversion), and 8 mentoring sessions for supportive transition to options for alternative income (HIVRR+S+FLM) (n=330).*

*Revision note: Following COVID-19, with approval from NIMH (on record if requested), the HIVRR+S+FLM treatment of the study has been combined with the HIVRR+S+FL treatment arm. The total sample size has been revised to 542 participants, with approval from NIMH. Moreover, biomarker data collection at 6 and 12 months were suspended due to COVID-19.

DETAILED DESCRIPTION:
Female Sex Workers (FSWs) in sub-Saharan Africa (SSA) have been identified as a high-risk group for the spread of HIV/AIDS, with those in poor areas and "HIV hotspots" being especially vulnerable. Research has shown that the primary reason poor women engage in commercial sex work is financial instability. Given these challenges, poor women require support over and above HIV prevention education. We propose to test the impact of adding economic empowerment (EE) components to traditional HIV risk reduction (HIVRR) to reduce new incidence of sexually transmitted infections (STIs) and of HIV among FSWs in Rakai and Masaka districts in Uganda. Guided by social-cognitive and asset theories, the study provides an avenue for FSWs to explore alternative means of safe and sustainable income to replace sex work. The study is informed by a previously tested microfinance (MF) intervention for FSWs in Mongolia, a pilot study conducted with FSWs in Masaka and Rakai, surveillance studies by RHSP, and EE interventions among AIDS-affected families in Uganda. Using a cluster-design we will randomly assign 990 FSWs from 33 matched town centers to one of three study arms (11 town centers in each condition): (1) A control arm comprising of treatment as usual (TAU) for FSWs in the study area bolstered with 4 evidence-based sessions of HIVRR provided by local providers (n=330); or (2) A treatment arm including TAU, 4 sessions of HIVRR, combined with receipt of a matched savings account (HIVRR+S+FL) to be used on short- and/or long-term consumption and skills development as per participants' own discretion plus 6 sessions of financial literacy (n=330); or (3) A treatment arm including TAU, 4 sessions of HIVRR, combined with a matched savings account to be used on short-term and/or long term consumption and skills development as per a participant's own discretion plus 6 sessions of financial literacy and 8 mentoring sessions for supportive transition to alternative income options (HIVRR+S+FLM) (n=330).* This RCT study's aims are to:

Aim1: Examine the impact of a financial savings-led MF intervention using HIVRR+S+FL and HIVRR+S+FLM on HIV biological and behavioral outcomes in FSWs (Primary outcomes: women's cumulative incidence of biologically confirmed STIs and reported number and proportion of unprotected sexual acts with regular and paying partners; Secondary outcomes: women's rate of new HIV cases, proportion of monthly income from sex and nonsex work, reported number and proportion on preventive behaviors, and for HIV+ women only, viral load as a marker of ART adherence).

Aim 2: Examine intervention mediation and effect modification to assess whether primary outcomes are mediated/moderated by participant characteristics; whether key theory-driven variables and Behavioral Economics measures mediate/moderate intervention outcomes.

Aim 3: Qualitatively and quantitatively examine implementation in each study condition; Aim 4: Assess the cost and cost-effectiveness of the HIVRR+S+FL and HIVRR+S+FLM intervention compared with traditional HIVRR in terms of cumulative number of STI and HIV cases averted over the 24-month period.

*Revision note: Following COVID-19, with approval from NIMH (on record if requested), the HIVRR+S+FLM treatment of the study has been combined with the HIVRR+S+FL treatment arm. The total sample size has been revised to 542 participants, with approval from NIMH. Moreover, biomarker data collection at 6 and 12 months were suspended due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years old
2. report having engaged in vaginal or anal intercourse in the past 90 days in exchange for money, alcohol, or other goods
3. report at least one episode of unprotected sexual intercourse in the past 90 days with either a paying, casual, or regular sexual partner.

Exclusion Criteria:

1. have a cognitive or severe psychiatric impairment that would prevent comprehension of study procedures as assessed during Informed Consent process
2. are unwilling or unable to commit to completing the study
3. have previously been randomized.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be female.
Enrollment: 542 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Ssewamala, PhD, Principal Investigator — Washington University School of Medicine; Susan Witte, PhD, Principal Investigator — Columbia University
Locations (1):
- International Center for Child Health and Development Field Office, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PIs and indicates the data will be used for the purposes of research (per CFR Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Brown School of Social Work and Columbia University School of Social Work Office of Sponsored Projects' data sharing agreements.

REFERENCES:
- [Derived] Witte SS, Ssewamala FM, Kiyingi J, Bellamy SL, Yang LS, Nabunya P, Bahar OS, Mayo-Wilson LJ, Tozan Y, Mwebembezi A, Kagaayi J. A cluster-randomized controlled trial of a combination HIV risk reduction and economic empowerment intervention for women engaged in sex work in Uganda. J Int AIDS Soc. 2025 Nov;28(11):e70057. doi: 10.1002/jia2.70057. PMID 41211615
- [Derived] Nabayinda J, Witte SS, Kizito S, Nanteza F, Nsubuga E, Sensoy Bahar O, Nabunya P, Ssewamala FM. The impact of an economic empowerment intervention on intimate partner violence among women engaged in sex work in southern Uganda: A cluster randomized control trial. Soc Sci Med. 2024 May;348:116846. doi: 10.1016/j.socscimed.2024.116846. Epub 2024 Apr 3. PMID 38581814
- [Derived] Sensoy Bahar O, Nabunya P, Nabayinda J, Witte S, Kiyingi J, Nsubuga E, Schriger S, Nattabi J, Mayo-Wilson LJ, Nakigudde J, Tozan Y, Ssewamala FM. "I decided in my heart I have to complete the sessions": A qualitative study on the acceptability of an evidence-based HIV risk reduction intervention among women engaged in sex work in Uganda. PLoS One. 2023 Jan 12;18(1):e0280138. doi: 10.1371/journal.pone.0280138. eCollection 2023. PMID 36634037
- [Derived] Jennings Mayo-Wilson L, Yen BJ, Nabunya P, Bahar OS, Wright BN, Kiyingi J, Filippone PL, Mwebembezi A, Kagaayi J, Tozan Y, Nabayinda J, Witte SS, Ssewamala FM. Economic Abuse and Care-seeking Practices for HIV and Financial Support Services in Women Employed by Sex Work: A Cross-Sectional Baseline Assessment of a Clinical Trial Cohort in Uganda. J Interpers Violence. 2023 Jan;38(1-2):NP1920-NP1949. doi: 10.1177/08862605221093680. Epub 2022 May 5. PMID 35510547
- [Derived] Witte SS, Filippone P, Ssewamala FM, Nabunya P, Bahar OS, Mayo-Wilson LJ, Namuwonge F, Damulira C, Tozan Y, Kiyingi J, Nabayinda J, Mwebembezi A, Kagaayi J, McKay M. PrEP acceptability and initiation among women engaged in sex work in Uganda: Implications for HIV prevention. EClinicalMedicine. 2022 Jan 28;44:101278. doi: 10.1016/j.eclinm.2022.101278. eCollection 2022 Feb. PMID 35128367
- [Derived] Nabunya P, Kiyingi J, Witte SS, Sensoy Bahar O, Jennings Mayo-Wilson L, Tozan Y, Nabayinda J, Mwebembezi A, Tumwesige W, Mukasa B, Namirembe R, Kagaayi J, Nakigudde J, McKay MM, Ssewamala FM. Working with economically vulnerable women engaged in sex work: Collaborating with community stakeholders in Southern Uganda. Glob Public Health. 2022 Jul;17(7):1215-1231. doi: 10.1080/17441692.2021.1916054. Epub 2021 Apr 21. PMID 33881949
- [Derived] Ssewamala FM, Sensoy Bahar O, Tozan Y, Nabunya P, Mayo-Wilson LJ, Kiyingi J, Kagaayi J, Bellamy S, McKay MM, Witte SS. A combination intervention addressing sexual risk-taking behaviors among vulnerable women in Uganda: study protocol for a cluster randomized clinical trial. BMC Womens Health. 2019 Aug 17;19(1):111. doi: 10.1186/s12905-019-0807-1. PMID 31419968

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following COVID-19, with approval from NIMH (on record if requested), the HIVRR+S+FLM treatment arm of the study has been combined with the HIVRR+S+FL treatment arm. The total sample size has been revised to 542 participants, with approval from NIMH.
Groups:
- Control Arm: Bolstered Treatment: Women in the control condition received treatment as usual (TAU) which includes: health education, HIV testing services, STI screening and treatment in a 2-hour session, provided on a quarterly basis. TAU was bolstered with 4 sessions of an evidence-based, HIV/STI risk reduction (HIVRR) intervention
- Treatment Arm: HIVRR+S+FL: Women in this arm received TAU and the 4 HIVRR sessions, plus two additional intervention components: 1) Financial Literacy: This evidence-based Financial Education Core Curriculum addresses the importance of savings, banking services, budgeting debt management; and 2) Matched savings individual development account.The accounts introduce women to financial management skills, introduce them to formal financial institutions, and by matching their deposits, incentivize women to save small amounts. Each woman received an IDA held in their own name. Women were allowed to contribute up to 50,000 shillings (~15 USD) per month towards their IDAs. The maximum amount of women's contribution was an equivalent of US$15 per month for 10 months. During the intervention, monthly account statements were generated for women to note their accumulated savings. During the intervention, women had direct access to both their personal savings deposited in the accounts and the match provided by the study. Women's monthly transactions were tracked using financial diaries.
Period: Overall Study
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Started | 186 | 356
Completed | 155 | 291
Not Completed | 31 | 65
Not completed — Lost to Follow-up | 31 | 65

BASELINE CHARACTERISTICS:
Groups:
- Control Arm: Bolstered Treatment: Women in the control condition (and in the treatment arms) will receive treatment as usual (TAU) which includes: health education, HIV testing services, STI screening and treatment in a session that lasts about 2 hours, provided on a quarterly basis. This will be bolstered with 4 sessions of an evidence-based, HIV/STI risk reduction (HIVRR) intervention
- Treatment Arm: HIVRR+S+FL: Women in this arm will receive TAU for FSW and the 4 HIVRR sessions, and two additional intervention components: 1) Financial Literacy: This evidence-based Financial Education Core Curriculum addresses the importance of savings, banking services, budgeting debt management; and 2) Matched savings individual development account.The accounts introduce women to financial management skills, introduce them to formal financial institutions, and by matching their deposits, incentivize women to save small amounts. Each woman will receive an IDA held in her own name. Women will be allowed and indeed encouraged to contribute up to 50,000 shillings (~15 USD) per month towards their IDAs. The maximum amount of women's contribution to be matched will be an equivalent of US$15 per month for 10 months. During the intervention, monthly account statements will be generated for women to note their accumulated savings. During the intervention, women will have direct access to both their personal savings deposited in the accounts and the match provided by the study.
- Total: Total of all reporting groups
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL | Total
Number analyzed (Participants) | 186 | 356 | 542
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (7.18) | 31.4 (7.39) | 31.4 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 356 | 542
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 186 | 356 | 542
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 186 | 356 | 542
Number of Participants with STIs [Number; unit: participants] — Number of participants testing positive for any of the three STIs including Gonorrhea, Trichomonas or Chlamydia, assessed using biomarkers.
  participants | 24 | 33 | 57
Number of Participants with HIV [Number; unit: participants] — Number of participants testing positive for HIV assessed using biomarker data.
  participants | 79 | 141 | 220
Number of Unprotected Sexual Acts with a Regular Partner [Mean (Standard Deviation); unit: unprotected sexual acts] — Number of unprotected sexual acts (e.g. vaginal and anal sexual acts) with a regular partner.
  unprotected sexual acts | 3.96 (8.96) | 4.52 (9.41) | 4.33 (9.26)
Number of Unprotected Sexual Acts with a Paying Partner [Mean (Standard Deviation); unit: unprotected sexual acts] — Number of unprotected sexual acts (e.g. vaginal and anal sexual acts) with a paying partner
  unprotected sexual acts | 3.09 (11.83) | 2.41 (8.86) | 2.64 (9.98)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With STIs
Description: Number of participants testing positive for any of the three STI including Gonorrhea, Trichomonas or Chlamydia, as assessed using biomarkers
Time Frame: 24 months
Population: Due to missing data, the number of participants analyzed reduced to 411 (35 participants missing STI data).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 143 | 268
Participants | 17 | 39

2. Primary Outcome: Number of Unprotected Sexual Acts With a Regular Partner
Description: Number of unprotected sexual acts (e.g. vaginal and anal sexual acts) with a regular partner
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: unprotected sexual acts
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 155 | 291
unprotected sexual acts | 5.16 (8.25) | 4.39 (8.52)

3. Primary Outcome: Number of Unprotected Sexual Acts With a Paying Partner
Description: Number of unprotected sexual acts (e.g. vaginal and anal sexual acts) with a paying partner
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: unprotected sexual acts
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 155 | 291
unprotected sexual acts | 0.45 (1.23) | 0.62 (1.87)

4. Secondary Outcome: Number of Participants With HIV
Description: Number of participants testing positive for HIV, assessed using biomarker data.
Time Frame: 24 months
Population: Only participants who tested HIV negative as 18 months follow-up assessments were retested.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 155 | 291
Participants | 65 | 117

5. Secondary Outcome: Viral Suppression
Description: Viral Suppression for women living with HIV was assessed using detectable vs undetectable viral load.
Time Frame: 24 months
Population: Viral suppression was only assessed from participants who tested positive for HIV at 24-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 65 | 117
Participants | 50 | 91

6. Secondary Outcome: Proportion of Income From Sex Work
Description: Participants reported their average total income and proportion of income from sex work. Proportion of income from sex work was calculated as average monthly total income as the denominator and income from sex work as the numerator.
Time Frame: 24 months
Measure: Median (Full Range); unit: proportion of income
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 155 | 291
proportion of income | 0.57 [0.40 to 0.80] | 0.58 [0.33 to 1]

7. Secondary Outcome: Preventive Behaviors/Condom Use With a Paying Partner
Description: Preventive behaviors was assessed by number of times a participant used condoms with a paying partner during sexual acts.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: preventive behaviors
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 155 | 291
preventive behaviors | 2.12 (2.99) | 1.89 (2.51)

8. Secondary Outcome: Preventive Behaviors/Condom Use With a Regular Partner
Description: Preventive behaviors was assessed by number of times a participant used condoms with a regular partner during sexual acts.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: preventive behaviors
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
Number analyzed (Participants) | 155 | 291
preventive behaviors | 0.41 (2.15) | 0.34 (1.53)

ADVERSE EVENTS:
Time Frame: 24-months
Arm/Group | Control Arm: Bolstered Treatment | Treatment Arm: HIVRR+S+FL
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/356
Serious Adverse Events (participants affected / at risk) | 0/186 | 0/356
Other Adverse Events (participants affected / at risk) | 0/186 | 0/356

LIMITATIONS AND CAVEATS:
Study implementation (including recruitment, data collection and intervention delivery) was greatly impacted by COVID-19 and associated mitigating risks. Following COVID-19, with approval from NIMH (on record if requested), the HIVRR+S+FLM treatment arm of the study was combined with the HIVRR+S+FL treatment arm. The total sample size was revised to 542 participants, with approval from NIMH. Moreover, biomarker data collection at 6 and 12 months were suspended due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT03583541/Prot_SAP_000.pdf